CLINICAL TRIAL: NCT04409080
Title: A Phase 1/2 Study of REGN7257 (Anti-Interleukin 2 Receptor Subunit Gamma [IL2RG] Monoclonal Antibody) in Patients With Severe Aplastic Anemia That Is Refractory to or Relapsed on Immunosuppressive Therapy
Brief Title: REGN7257 in Adult Patients With Severe Aplastic Anemia That Is Refractory to or Relapsed on Immunosuppressive Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R7257-RAA-1947; 2020-002031-29 (EudraCT Number); 2023-508601-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-08

CONDITIONS: Severe Aplastic Anemia (SAA)
Keywords: Immunosuppressive therapy (IST); Refractory; Relapsed
MeSH Terms: conditions — Anemia, Aplastic; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A: Single ascending dose (SAD) escalation cohorts
  Interventions: Drug: REGN7257
- Part B (Experimental): Part B: Multiple REGN7257 dosages.
  Interventions: Drug: REGN7257

INTERVENTIONS:
Drug: REGN7257 — Administered by intravenous (IV) infusion, in Part A and B.

SUMMARY:
This study is researching an experimental drug called REGN7257 (called "study drug"). The study is focused on patients who have severe aplastic anemia (SAA), a disease of the bone marrow resulting in an impairment of the production of blood cells.

The main purpose of this two-part study (Part A and Part B) is to test how safe and tolerable REGN7257 is in patients with SAA in which other Immunosuppressive therapies (ISTs) have not worked well.

The study is looking at several other research questions to better understand the following properties of REGN7257:

* Side effects that may be experienced by participants taking REGN7257
* How REGN7257 works in the body
* How much REGN7257 is present in blood after dosing
* If REGN7257 works to raise levels of certain blood counts after treatment
* How quickly REGN7257 works to raise levels of certain blood counts
* In patients for whom REGN7257 works to raise levels of certain blood counts after treatment, how many continue to show such a response throughout the study
* If REGN7257 works to lower the number of platelet and red blood cell transfusions needed
* How REGN7257 changes immune cell counts and composition
* How the body reacts to REGN7257 and if it produces proteins that bind to REGN7257 (this would be called the formation of anti-drug antibodies [ADA])

DETAILED DESCRIPTION:
The trial was intended to be a Phase 1/2 trial, but no participants were enrolled in Phase 2

ELIGIBILITY:
Key Inclusion Criteria:

1. Part A: SAA that is IST-refractory or IST-relapsed, as defined in the protocol
2. Part B: SAA that is IST-relapsed, as defined in the protocol
3. Hematopoietic stem cell transplantation (HSCT) is not available or suitable as a treatment option or has been refused by the patient
4. Adequate hepatic and renal function as defined in the protocol

Key Exclusion Criteria:

1. Diagnosis of Fanconi anemia or other congenital bone marrow failure syndrome as defined in the protocol
2. Evidence of myelodysplastic syndrome as defined in the protocol
3. Paroxysmal nocturnal hemoglobinuria (PNH) with evidence of clinically significant hemolysis (eg, treatment indicated) or history of PNH-associated thrombosis
4. Treatment with a T cell-depleting agent (eg, ATG or alemtuzumab) within 6 months prior to dosing
5. Treatment with a calcineurin inhibitor (eg, cyclosporine) within 4 weeks prior to dosing for patients enrolled in Part A
6. Treatment with eltrombopag or investigational thrombopoietin receptor agonist, Granulocyte Colony-Stimulating Factor (G-CSF), or an androgen (eg, danazol), within 2 weeks prior to dosing
7. HIV, hepatitis B or hepatitis C positive by serological testing at the screening visit as defined in the protocol
8. Active tuberculosis, latent tuberculosis infection (LTBI) or history incompletely-treated tuberculosis or LTBI
9. Active infection as defined in the protocol

Note: Other protocol-defined inclusion/ exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 12 months post-treatment, approximately 52 weeks
  Part A
Incidence of serious adverse events (SAEs) | 12 months post-treatment, approximately 52 weeks
  Part A
Incidence and severity of treatment-emergent adverse events (TEAEs) | 12 months post-treatment, approximately 52 weeks
  Part A
Incidence of serious adverse events (SAEs) | Through the end of study visit, approximately 78 weeks
  Part B
Incidence and severity of treatment-emergent adverse events (TEAEs) | Through the end of study visit, approximately 78 weeks
  Part B
Overall response rate (ORR) | At 6 months, approximately 26 weeks
  Part B

SECONDARY OUTCOMES:
ORR | At 3 months, approximately 12 weeks
  Parts A and B
Complete response (CR) | At 3 months, approximately 12 weeks
  Parts A and B
Partial response (PR) | At 3 months, approximately 12 weeks
  Parts A and B
Time to best response | Up to 12 months
  Part A
Time to best response | Up to 18 months
  Part B
Time to first response | Up to 12 months
  Part A
Time to first response | Up to 18 months
  Part B
Any clinical response | Until the end of study, approximately week 52
  Part A
Any clinical response | Until the end of study, approximately week 78
  Part B
Platelet transfusions per month over time | Up to 12 months
  Part A
Platelet transfusions per month over time | Up to 18 months
  Part B
Red blood cell transfusions per month over time | Up to 12 months
  Part A
Red blood cell transfusions per month over time | Up to 18 months
  Part B
Changes in lymphocyte cell counts | Up to 12 months
  Part A
Changes in lymphocyte cell counts | Up to 18 months
  Part B
Changes in neutrophil cell counts | Up to 12 months
  Part A
Changes in neutrophil cell counts | Up to 18 months
  Part B
Changes in hemoglobin cell counts | Up to 12 months
  Part A
Changes in hemoglobin cell counts | Up to 18 months
  Part B
Changes in reticulocyte cell counts | Up to 12 months
  Part A
Changes in reticulocyte cell counts | Up to 18 months
  Part B
Changes in platelet cell counts | Up to 12 months
  Part A
Changes in platelet cell counts | Up to 18 months
  Part B
Changes in the whole blood immune cell subsets (T cells) | Up to 12 months
  Part A
Changes in the whole blood immune cell subsets (T cells) | Up to 18 months
  Part B
Changes in the whole blood immune cell subsets (B cells) | Up to 12 months
  Part A
Changes in the whole blood immune cell subsets (B cells) | Up to 18 months
  Part B
Changes in the whole blood immune cell subsets [Natural killer (NK) cells] | Up to 12 months
  Part A
Changes in the whole blood immune cell subsets (NK cells) | Up to 18 months
  Part B
Drug concentrations in serum over time | Up to 12 months
  Part A
Drug concentrations in serum over time | Up to 18 months
  Part B
Incidence of treatment-emergent anti-drug antibody (ADA) over time | Up to 12 months
  Part A
Incidence of treatment-emergent ADA over time | Up to 18 months
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Hopital Saint-Louis - APHP, Paris, Île-de-France Region, France
- South Korea (5):
  - Gachon University Gil Hospital, Incheon, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul Capital Area
  - Samsung Medical Center, Seoul, Seoul Capital Area
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul, Seoul Capital Area
  - Ewha Womans University Medical Centre, Seoul, Seoul Capital Area
- United Kingdom (2):
  - St James's University Hospital, Leeds, West Yorkshire
  - King's College Hospital, London, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/